CLINICAL TRIAL: NCT04038814
Title: The Effectiveness of the Modified Bundle in the Prevention of Ventilator-associated Pneumonia in Adult Patients in the Intensive Care Unit.
Brief Title: The Effectiveness of the Modified Bundle in the Prevention of VAP.
Acronym: VAP
Status: Completed | Type: Observational
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, JAROSLAW PAWLIK, MD, Specialist of anaesthesiology and intensive care, An assistant of The Faculty of Medicine and Health Sciences, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: AFMKrakowU
Record Dates: First submitted 2019-07-27; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: VAP - Ventilator Associated Pneumonia
Keywords: VAP; Evac Endotracheal Tube with TaperGuard Cuff; MDR - multi drug resistant pathogens; SSD - subglottic secretion drainage,
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VAP1 - historical group: Routine prevention of VAP
  Interventions: Procedure: Routine prevention of VAP
- VAP2 - study group: Modified prevention of VAP
  Interventions: Procedure: Modified prevention of VAP

INTERVENTIONS:
Procedure: Routine prevention of VAP — Enhanced hand hygiene protocol, tube cuff pressure monitoring ( set on 25-30 mm Hg) every 12 hours and every time when we suspected under or over distention, fast withdrawal of sedation, moderate supportive mechanical ventilation ( tidal volume (VT) 5-8 ml/kg ideal body weight (IBW), positive end expiratory pressure (PEEP) 3-5 cmH2O, Plateau pressure (Ppl) < 25 cm H2O, normocapnia ), Proton Pump Inhibitors (PPIs) reduction, Selective oral decontamination (SOD) every 8 hours - 0,2% chlorhexidine digluconate mouthwash, Closed Tracheal Suction System (CTSS) - changed every 7 day, 30-45% lifting of the thorax
  Groups: VAP1 - historical group
Procedure: Modified prevention of VAP — 3 modifications of the routine bundle in the prevention of VAP:
  * Endotracheal tube ( Shiley Evac Endotracheal tube with TaperGuard Cuff) and tracheostomy tubes (Tracheostomy Tube Cuffed Seal Guard) instead of regular tubes,
  * Automatic, continuous tube cuff pressure monitoring ( Covidien Shiley M Pressure Control Automatic Cuff Controller ( 25-30 mmHg),
  * Automatic continuous subglottic secretion drainage
  Groups: VAP2 - study group

SUMMARY:
Ventilator-associated pneumonia (VAP) is an important cause of prolonged intensive care unit and hospital length of stay, healthcare costs and mortality in mechanically ventilated patients. There are an international guidelines for VAP diagnosis, treatment and prevention (Infectious Diseases Society of America(IDSA)/American Thoracic Society (ATS) 2016 and European Respiratory Society (ERS) / European Society of Intensive Care Medicine (ESICM) / European Society of Clinical Microbiology and Infectiuos Diseases (ESCMID) / Asociacion Latinoamericana del Torax (ALAT) 2017) routinely used in most ICUs. The investigator planed on comparing two strategies for prevention of VAP in mechanically ventilated patients: the routine VAP bundle ( historical group - VAP1) and the modified VAP bundle ( study group - VAP2) by using 3 modifications ( Shiley Evac Endotracheal tube with TaperGuard Cuff, Automatic continuous subglottic secretion drainage (SSD) and continuous tube cuff pressure monitoring).

The aim of the study is an assessment of the effectiveness of the modified prevention of VAP in reduction of: early and late VAP cases, mechanical ventilation days (MV), length of stay (LOS) in the ICU, 28 day mortality and multi drug resistent pathogens (MDR) cases in adult ICU patients.

ELIGIBILITY:
Inclusion Criteria:

VAP2 - study group

* mechanically ventilated patients with an artificial airways (endotracheal tube, tracheostomy tube)
* age over 18 years
* modified bundle in the prevention of VAP

VAP1 - historical group

* mechanically ventilated patients with an artificial airways (endotracheal tube, tracheostomy tube)
* patients hospitalised in the ICU for last 12 months before modified bundle in the prevention of VAP has been started (from 01.05.2017 to 30.04.2018)
* age over 18 years
* routine bundle in the prevention of VAP

Exclusion Criteria:

* lack of an informed consent in awake patients in the ICU
* age under 18 years
* patients with no mechanical ventilation in the ICU
* patients with probability of mechanical ventilation days and LOS in the ICU less than 48 hours
* patients intubated and mechanically ventilated without the bundle in the prevention of VAP for a period of time longer than 12 hours before the admission to the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group were male and female patients ( neurosurgical, cardiological, general surgical and non cardiological internal medicine type) in adult ICU. Each enrolled patient was mechanically ventilated for a period longer than 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Early VAP | day: 2 - 5 of mechanical ventilation
  Total VAP cases in the ICU ( CEPPIS /Chest Echocardiography and Procalcitonin Pulmonary Infection Score/ criteria ) with early beginning of the pneumonia symptoms.
Late VAP | day: 6 - the last day in ICU
  total VAP cases in the ICU ( CEPPIS criteria ) with late beginning of the pneumonia symptoms

SECONDARY OUTCOMES:
LOS | day: 1 - the last day in the ICU, but at least 2 days
  lenght of stay in the ICU (days)
MV | day: 1 - the last day in the ICU, but at least 2 days
  Duration of mechanical ventilation (days) in the ICU
nonMV | day: 1 - the last day in the ICU,
  Total non mechanical ventilation days in the ICU
Mortality | day: 1 - 28
  Mortality of adult mechanically ventilated patients in the ICU
MDR | day: 1 - the last day in the ICU,
  Number of cases with multi drug resistant (MDR) pathogens detected in specimens of mucus taken from the lower airways in mechanically ventilated patients in the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: JAROSLAW PAWLIK, MD, Principal Investigator — Andrzej Frycz Modrzewski Krakow University
Locations (1):
- Anaesthesiology and Intensive Care Unit St. Raphael Hospital, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided